CLINICAL TRIAL: NCT05741164
Title: Impact of Beta-2 Adrenergic Blockade With Checkpoint Inhibition in Checkpoint Inhibitor Refractory Metastatic Triple Negative Breast Cancer
Brief Title: Propranolol and Pembrolizumab for Tumor Re-sensitization and Treatment of Patients With Checkpoint Inhibitor Refractory Metastatic or Unresectable Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 2612022; NCI-2023-00641 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 2612022 (Other: Roswell Park Cancer Institute); K08CA279766 (NIH)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma; Refractory Triple-Negative Breast Carcinoma; Unresectable Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy; Specimen Handling; pembrolizumab; Propranolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (propranolol and pembrolizumab) (Experimental): Patients receive propranolol PO and pembrolizumab IV while on study. Patients undergo CT scan, blood sample collection and may undergo tumor biopsy during screening and on study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Pembrolizumab; Drug: Propranolol; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Propranolol — Given PO
  Other Names: 1-[(1-Methylethyl)amino]-3-(1-naphthalenyloxy)-2-propanol
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well propranolol and pembrolizumab work to cause tumor re-sensitization and therefore treatment in patients with triple negative breast cancer that has not responded to previous checkpoint inhibitor therapy (refractory), cannot be removed by surgery (unresectable) or has spread from where it first started (primary site) to other places in the body (metastatic). Propranolol is a drug that is classified as a beta-blocker. Beta-blockers affect the heart and circulation. Beta-blockers, like propranolol, may help to counteract effects of certain stress hormones produced by the body during cancer treatment and may increase the effectiveness of the pembrolizumab. Pembrolizumab is a drug that is classified as an immune checkpoint inhibitor. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Propranolol may be able to re-sensitize the cells of the immune system to respond to the checkpoint inhibitor pembrolizumab in patients with checkpoint inhibitor refractory metastatic or unresectable triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the efficacy of propranolol on tumor re-sensitization, when given in combination with pembrolizumab in patients with checkpoint inhibitor refractory metastatic triple negative breast cancer.

SECONDARY OBJECTIVES:

I. Assess 6-month progression-free and overall survival per immune-related Response Evaluation Criteria in Solid Tumors (irRECIST).

II. Safety and tolerability of propranolol when given in combination with pembrolizumab.

EXPLORATORY OBJECTIVES:

I. Assess changes in immune markers (pre-treatment versus [vs] post-treatment) in biopsy and peripheral blood.

II. Correlate perceived stress scale with immune exhaustion markers and immune cells in the peripheral blood and tumor.

OUTLINE: Patients receive propranolol orally (PO) and pembrolizumab intravenously (IV) while on study. Patients undergo computed tomography (CT) scan, blood sample collection and may undergo tumor biopsy during screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Have pathologically confirmed diagnosis of unresectable or metastatic triple negative breast cancer (TNBC) with no curative treatment options
* No chemotherapy, radiotherapy, or major surgery within 4 weeks of protocol treatment
* Checkpoint inhibitor refractory patients (i.e., no longer responding to chemotherapy and checkpoint inhibitor) who have disease progression on prior line of chemotherapy and pembrolizumab, and, who in the opinion of the physician, can continue checkpoint inhibitor
* Patients must be agreeable to pre- and 6-week post treatment biopsy in part 1 of the study

  * The pre-treatment biopsy for this study must be taken at least 4 weeks after all previous chemotherapy (pembrolizumab is allowed during this period)
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g. hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of =< 1
* Platelets >= 100,000/uL
* Hemoglobin >= 9.0 g/dL
* Absolute neutrophil count (ANC) >= 1500/uL
* Total bilirubin =< institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional ULN
* Creatinine clearance >= 50 mL/min per Cockcroft-Gault equation
* HbA1C <=8.5
* Have measurable disease per RECIST 1.1 criteria present
* Ability to swallow and retain oral medication
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients currently treated with systemic immunosuppressive agents, including steroids, are ineligible until 3 weeks after removal from immunosuppressive treatment
* Patients with active autoimmune disease, requiring ongoing immunosuppressive therapy or history of transplantation
* Patients with rapidly progressive disease/ symptomatic disease
* Patients with primary resistance (i.e., did not respond to initial treatment with chemotherapy plus checkpoint inhibitor) with progressive disease at 12 weeks after starting chemotherapy and pembrolizumab
* Patients who are pregnant or nursing. Women of childbearing potential (WOCBP) will have to undergo a urine pregnancy test as part of screening
* Participants with symptomatic known brain metastases < 4 weeks from radiation treatment should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of malignancy other than breast cancer within 5 years prior to screening, with the exception of those with a negligible risk of metastases or death
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Unwilling or unable to follow protocol requirements
* Contraindications to the use of beta-blockers, like: uncontrolled depression, unstable angina pectoris, uncontrolled heart failure (grade III or IV), hypotension (systolic blood pressure < 100 mmHg), severe asthma or chronic obstructive pulmonary disease (COPD), uncontrolled type I or type II diabetes mellitus (hemoglobin A1C [HbA1C] > 8.5 or fasting plasma glucose > 160 mg/dl at screening), symptomatic peripheral arterial disease or Raynaud's syndrome, untreated pheochromocytoma, current use of beta-blockers or non-dihydropyridine calcium channel blockers
* Any additional condition which in the investigator's opinion deems the participant an unsuitable candidate to receive the study drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Objective response | Up to 6 months
  Efficacy as determined by immune-related Response Evaluation Criteria in Solid Tumors (irRECIST). Will be summarized using frequencies and relative frequencies. The best response within the first 6 months will be determined as the best objective response.

SECONDARY OUTCOMES:
Progression free survival | The time treatment initiation until disease progression (per irRECIST), death due to any cause, subsequent therapies (treated as censored), or last follow-up, assessed up to 6 months
  This will be summarized using standard Kaplan-Meier methods with 90% confidence intervals obtained for the median and 6-month rates.
Overall survival | The time from treatment initiation until death due to any cause or last follow-up, assessed up to 6 months
  Measured per irRECIST. This will be summarized using standard Kaplan-Meier methods with 90% confidence intervals obtained for the median and 6-month rates.
Incidence of adverse events of propranolol when given in combination with pembrolizumab | Up to 2 years
  Toxicities and adverse events (as per Common Terminology Criteria for Adverse Events version 5.0) will be summarized by attribution and grade using frequencies and relative frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Sheheryar Kabraji, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States